CLINICAL TRIAL: NCT04557618
Title: Transcutaneous Auricular Vagus Nerve Stimulation Following Spontaneous Subarachnoid Hemorrhage
Brief Title: Auricular VNS Following Subarachnoid Hemorrhage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anna Huguenard (Other)
Responsible Party: Sponsor-Investigator, Anna Huguenard, Assistant Professor of Neurosurgery, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202007034
Record Dates: First submitted 2020-09-04; First posted 2020-09-21 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Subarachnoid Hemorrhage
Keywords: Vagal nerve stimulation
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either stimulation or sham stimulation arms
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All participants will be fitted with an auricular stimulator, but blinded to whether they are receiving stimulation or not. Outcome scores will be assessed and recorded by clinicians blinded to treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Auricular VNS Stimulation (Experimental): Participants receive twice daily auricular vagal nerve stimulation
  Interventions: Device: Auricular Vagus Nerve Stimulation
- Sham Auricular VNS Stimulation (Sham Comparator): Participants will have an auricular vagal nerve stimulator applied twice daily, without the stimulation applied
  Interventions: Device: Sham Auricular Vagus nerve Stimulation

INTERVENTIONS:
Device: Auricular Vagus Nerve Stimulation — Transcutaneous auricular vagal nerve stimulation
  Arms: Auricular VNS Stimulation
Device: Sham Auricular Vagus nerve Stimulation — Transcutaneous auricular vagal nerve ear clip applied without current
  Arms: Sham Auricular VNS Stimulation

SUMMARY:
This study will evaluate whether non-invasive auricular vagal nerve stimulation lowers inflammatory markers, and improves outcomes following spontaneous subarachnoid hemorrhage.

DETAILED DESCRIPTION:
Vagal nerve stimulation (VNS) has been studied in several inflammatory conditions, and has been implemented in animal models of subarachnoid hemorrhage (SAH) with promising results. The purpose of the proposed study is to determine how applying auricular VNS in patients presenting with spontaneous SAH impacts their expression of inflammatory markers in their blood and cerebrospinal fluid (CSF), and how it impacts their clinical course and outcomes.

This study will involve randomizing patients to stimulation with VNS, or sham stimulation. Blood and CSF will be collected on admission, and serially throughout the patient's admission. Clinical events tracked during the hospital stay include development of cerebral vasospasm, need for CSF diversion via a shunt, stress-induced cardiomyopathy, and development of stroke or global cerebral ischemia. Outcomes following admission will include functional scores at discharge, and at follow-up visits for up to 2 years after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous subarachnoid hemorrhage

Exclusion Criteria:

* Trauma-induced subarachnoid hemorrhage
* Ongoing chemotherapy
* Taking immunosuppressive medications for other medical illnesses
* Presence of a pacemaker
* Prolonged bradycardia at time of admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Inflammatory markers in the serum on admission | On hospital day 1
  TNF alpha from blood draw
Change in inflammatory markers in the serum | Through hospital admission, average of 4 weeks
  TNF alpha from blood draws
Inflammatory markers in the CSF on admission | On hospital day 1
  TNF alpha from cerebrospinal fluid
Change in inflammatory markers in the CSF | Through hospital admission, average of 4 weeks
  TNF alpha from cerebrospinal fluid
Cerebral vasospasm | Through hospital admission, average of 4 weeks
  Presence of moderate/severe radiographic vasospasm
Hydrocephalus | Through hospital admission, average of 4 weeks
  Need for permanent CSF diversion via a ventricular shunt

SECONDARY OUTCOMES:
Inflammatory markers in the serum on admission | On hospital day 1
  IL-12, GM-CSF, IFN gamma, IL-1b, IL-10, IL-13, IL-17A, IL-2, IL-4, IL-5, IL-6, IL-8from blood draws
Change in inflammatory markers in the serum | Through hospital admission, average of 4 weeks
  IL-12, GM-CSF, IFN gamma, IL-1b, IL-10, IL-13, IL-17A, IL-2, IL-4, IL-5, IL-6, IL-8 from blood draws
Inflammatory markers in the CSF on admission | On hospital day 1
  IL-12, GM-CSF, IFN gamma, IL-1b, IL-10, IL-13, IL-17A, IL-2, IL-4, IL-5, IL-6, IL-8, from cerebrospinal fluid
Change in inflammatory markers in the CSF | Through hospital admission, average of 4 weeks
  IL-12, GM-CSF, IFN gamma, IL-1b, IL-10, IL-13, IL-17A, IL-2, IL-4, IL-5, IL-6, IL-8, from cerebrospinal fluid
Cerebral vasospasm | Through hospital admission, average of 4 weeks
  Additional features of vasospasm: 1) Number of vascular studies obtained, 2) Need for blood pressure augmentation or hypervolemia, 3) Need for intraarterial or intrathecal vasodilator, 4) Need for angioplasty
Cerebral ischemia | Through hospital admission, average of 4 weeks
  Presence of cerebral ischemia based on the following criteria: Radiographic evidence of a new infarct or stroke
Hydrocephalus | Through hospital admission, average of 4 weeks
  Duration of temporary CSF diversion via an external ventricular drain
Clinical outcome | 2 years
  Modified Rankin Scale for Neurological Disability (minimum score 0, maximum score 6, better outcomes have lower scores)
Stressed-induced cardiomyopathy | Through hospital admission, average of 4 weeks
  Presence of stressed-induced cardiomyopathy based on any of the following criteria: 1) New troponin elevation, 2) New EKG changes (specifically ST segment elevation, ST segment depression, left bundle branch block, prolonged QT interval), 3) New findings of cardiomyopathy on echocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Eric C Leuthardt, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tan G, Huguenard AL, Donovan KM, Demarest P, Liu X, Li Z, Adamek M, Lavine K, Vellimana AK, Kummer TT, Osbun JW, Zipfel GJ, Brunner P, Leuthardt EC. The effect of transcutaneous auricular vagus nerve stimulation on cardiovascular function in subarachnoid hemorrhage patients: A randomized trial. Elife. 2025 Jan 9;13:RP100088. doi: 10.7554/eLife.100088. PMID 39786346
- [Derived] Huguenard A, Tan G, Johnson G, Adamek M, Coxon A, Kummer T, Osbun J, Vellimana A, Limbrick D Jr, Zipfel G, Brunner P, Leuthardt E. Non-invasive Auricular Vagus nerve stimulation for Subarachnoid Hemorrhage (NAVSaH): Protocol for a prospective, triple-blinded, randomized controlled trial. PLoS One. 2024 Aug 23;19(8):e0301154. doi: 10.1371/journal.pone.0301154. eCollection 2024. PMID 39178291
- [Derived] Huguenard AL, Tan G, Rivet DJ, Gao F, Johnson GW, Adamek M, Coxon AT, Kummer TT, Osbun JW, Vellimana AK, Limbrick DD, Zipfel GJ, Brunner P, Leuthardt EC. Auricular Vagus Nerve Stimulation Mitigates Inflammation and Vasospasm in Subarachnoid Hemorrhage: A Randomized Trial. medRxiv [Preprint]. 2024 May 1:2024.04.29.24306598. doi: 10.1101/2024.04.29.24306598. PMID 38746275
- [Derived] Tan G, Huguenard AL, Donovan KM, Demarest P, Liu X, Li Z, Adamek M, Lavine K, Vellimana AK, Kummer TT, Osbun JW, Zipfel GJ, Brunner P, Leuthardt EC. The effect of transcutaneous auricular vagus nerve stimulation on cardiovascular function in subarachnoid hemorrhage patients: a safety study. medRxiv [Preprint]. 2024 Sep 8:2024.04.03.24304759. doi: 10.1101/2024.04.03.24304759. PMID 38633771
- [Derived] Huguenard AL, Tan G, Johnson GW, Adamek M, Coxon AT, Kummer TT, Osbun JW, Vellimana AK, Limbrick DD Jr, Zipfel GJ, Brunner P, Leuthardt EC. Non-invasive Auricular Vagus nerve stimulation for Subarachnoid Hemorrhage (NAVSaH): Protocol for a prospective, triple-blinded, randomized controlled trial. medRxiv [Preprint]. 2024 Mar 19:2024.03.18.24304239. doi: 10.1101/2024.03.18.24304239. PMID 38562875